CLINICAL TRIAL: NCT04153435
Title: Calcium for Out-of-Hospital Cardiac Arrest - A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Calcium for Out-of-Hospital Cardiac Arrest
Acronym: COCA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lars Wiuff Andersen (Other)
Collaborators: Central Denmark Region (Other); University of Aarhus (Other)
Responsible Party: Sponsor-Investigator, Lars Wiuff Andersen, Associate Professor, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 00002; 2019-003387-46 (EudraCT Number)
Record Dates: First submitted 2019-11-03; First posted 2019-11-06 (Actual); Results first posted 2022-02-25 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Heart Arrest, Out-Of-Hospital
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest | interventions — Calcium Chloride; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Calcium (Experimental): The intervention will consist of 5 mmol (10 mL ampoule) of calcium chloride (CaCl2) administered intravenously or intraosseously immediately after the first dose of adrenaline and again after the second dose of adrenaline.
  Interventions: Drug: Calcium Chloride
- Placebo (Placebo Comparator): The placebo will consist of 10 mL of 9 mg/mL sodium chloride (NaCl, "normal saline") administered intravenously or intraosseously immediately after the first dose of adrenaline and again after the second dose of adrenaline.
  Interventions: Drug: Sodium chloride 0.9%

INTERVENTIONS:
Drug: Calcium Chloride — Calcium chloride 5 mmol
  Other Names: CaCl2
  Arms: Calcium
Drug: Sodium chloride 0.9% — Placebo
  Arms: Placebo

SUMMARY:
This is an investigator-initiated, multicenter, randomized, placebo-controlled, parallel group, double-blind, superiority trial of calcium during adult out-of-hospital cardiac arrest. 430 adult patients with out-of-hospital cardiac arrest receiving at least one dose of adrenaline will be enrolled. The primary outcome is sustained return of spontaneous circulation and key secondary outcomes include survival at 30 days and survival at 30 days with a favorable neurological outcome.

ELIGIBILITY:
Inclusion Criteria:

* Out-of-hospital cardiac arrest
* Age ≥ 18 years
* Received at least one dose of adrenaline

Exclusion Criteria:

* Traumatic cardiac arrest - including drowning and external asphyxia (e.g., hanging, strangulation, or foreign object airway obstruction)
* Known or strongly suspected pregnancy
* Prior enrollment in the trial
* Received adrenaline during cardiac arrest before arrival of prehospital personnel with the study drug
* Clinical indication for calcium administration during the cardiac arrest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 397 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2022-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lars W Andersen, Principal Investigator — Aarhus University Hospital
Locations (1):
- Prehospital Emergency Medical Services, Aarhus N, Central Jutland, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Six months after the publication of the last results, all deidentified individual patient data will be made available for data sharing. Procedures, including re-coding of key variables, will be put in place to allow for complete deidentification of the data. Data will be completely anonymized according to Danish law.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Six months after the publication of the last results
Access Criteria: Data will be available for any research purpose to all interested parties who have approval from an independent review committee and who have a methodological sound proposal as determined by the steering committee of the current trial. Only the methodological qualities and not the purpose or objective of the proposal will be considered.

REFERENCES:
- [Derived] Vallentin MF, Granfeldt A, Meilandt C, Povlsen AL, Sindberg B, Holmberg MJ, Iversen BN, Maerkedahl R, Mortensen LR, Nyboe R, Vandborg MP, Tarpgaard M, Runge C, Christiansen CF, Dissing TH, Terkelsen CJ, Christensen S, Kirkegaard H, Andersen LW. Effect of calcium vs. placebo on long-term outcomes in patients with out-of-hospital cardiac arrest. Resuscitation. 2022 Oct;179:21-24. doi: 10.1016/j.resuscitation.2022.07.034. Epub 2022 Jul 30. PMID 35917866
- [Derived] Vallentin MF, Granfeldt A, Meilandt C, Povlsen AL, Sindberg B, Holmberg MJ, Iversen BN, Maerkedahl R, Mortensen LR, Nyboe R, Vandborg MP, Tarpgaard M, Runge C, Christiansen CF, Dissing TH, Terkelsen CJ, Christensen S, Kirkegaard H, Andersen LW. Effect of Intravenous or Intraosseous Calcium vs Saline on Return of Spontaneous Circulation in Adults With Out-of-Hospital Cardiac Arrest: A Randomized Clinical Trial. JAMA. 2021 Dec 14;326(22):2268-2276. doi: 10.1001/jama.2021.20929. PMID 34847226
- See also: Trial website — http://www.cocatrial.dk

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Calcium | Placebo
Started | 197 | 200
Completed | 197 | 200
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients received the trial drug and meeting all inclusion criteria and none of the exclusion criteria.
Groups:
- Total: Total of all reporting groups
Arm/Group | Calcium | Placebo | Total
Number analyzed (Participants) | 193 | 198 | 391
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (14) | 69 (14) | 68 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 52 | 114
  Male | 131 | 146 | 277
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Sustained Return of Spontaneous Circulation
Description: Palpable pulses or other signs of circulation without a need for chest compressions lasting at least 20 minutes.
Time Frame: Before or after hospital arrival (up to 2 hours after the cardiac arrest)
Population: Patients were analyzed according to their randomized assignment. The analyses only included patients receiving the first dose of the trial drug and meeting all inclusion criteria and no exclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Calcium | Placebo
Number analyzed (Participants) | 193 | 198
Participants | 37 | 53

2. Secondary Outcome: Number of Participants With 30-day Survival
Time Frame: 30 days after the cardiac arrest
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Calcium | Placebo
Number analyzed (Participants) | 193 | 198
Participants | 10 | 18

3. Secondary Outcome: Number of Participants With 30-day Favorable Neurological Outcome
Description: Neurological outcome will be assessed with the modified Rankin Scale (mRS) which is a scale from 0 to 6 assessing neurological/functional outcomes after brain damage with higher scores indicating worse neurological/functional outcomes. The scale will will be dichotomized as favorable (mRS 0-3) vs. unfavorable (mRS 4-6).
Time Frame: 30 days after the cardiac arrest
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Calcium | Placebo
Number analyzed (Participants) | 193 | 198
Participants | 7 | 15

ADVERSE EVENTS:
Time Frame: 30 days
Description: Adverse events were not collected.
Arm/Group | Calcium | Placebo
All-Cause Mortality (participants affected / at risk) | 183/193 | 180/198
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-21): https://cdn.clinicaltrials.gov/large-docs/35/NCT04153435/Prot_SAP_000.pdf